CLINICAL TRIAL: NCT04966949
Title: Lateral Prostate Capsule Sparing Versus Nerve Sparing Robot-assisted Radical Cystectomy-orthotopic Ileal Neobladder for Bladder Cancer in the Male
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SysMU-RARC2
Record Dates: First submitted 2021-07-09; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral prostate capsule sparing group (Experimental): Patients will be preverved the lateral prostate capsule during the resection of bladder and prostate of the operation.
  Interventions: Procedure: lateral prostate capsule sparing or neurovascular bundles sparing
- nerve sparing group (Active Comparator): Patients will be preverved the neurovascular bundles during the resection of bladder and prostate of the operation.
  Interventions: Procedure: lateral prostate capsule sparing or neurovascular bundles sparing

INTERVENTIONS:
Procedure: lateral prostate capsule sparing or neurovascular bundles sparing — When resect the bladder and prostate, the lateral prostate capsule or neurovascular bundles will be preserved.

SUMMARY:
To compare the perioperative, functional, and oncologic outcomes between nerve sparing and lateral prostate capsule sparing robot-assisted radical cystectomy with orthotopic ileal neobladder in male patients with bladder cancer.

DETAILED DESCRIPTION:
This study will enroll male patients with bladder cancer who will undergo robot-assisted radical cystectomy with orthotopic ileal neobladder. The patients will be distributed into two comparable groups according to surgical procedures: nerve sparing group and lateral prostate capsule sparing group. Patient demographics and pathologic, perioperative, functional, and oncologic outcomes will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 18 or older.
2. Patients those who are diagnosed with urothelial carcinoma.
3. Patients those who are without tumour in the bladder neck or urethra, and prostate cancer was ruled out by MRI and serum T-PSA<2.5ng/ml.
4. Patients those who are capable of receiving radical cystectomy with orthotopic ileal neobladder.
5. Patients those who are able to cooperate and complete the follow-up.
6. Patients those who volunteer to participate in this study and sign the informed consens.

Exclusion Criteria:

1. Patients thsoe who are diagnosed distant metastasis before surgery.
2. Patients those who are diagnosed with other malignancies.
3. Patients those who had received pelvic radiotherapy or major pelvic operation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
day-time continence rate | 6 months
  Patients were considered continent when they required 0 or 1 safety pad during the day time
night-time continence rate | 6 months
  Patients were considered continent when they required 0 or 1 safety pad during the night.
postoperative sexual function | 6 months
  The sexual function are evaluated by the international index of erectile function-5 (IIEF-5).

SECONDARY OUTCOMES:
perioperative complication rate | 3 months
operative time | 24 hours
estimated blood loss | 24 hours
overall survival | 1 year
recurrence-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No